CLINICAL TRIAL: NCT07071298
Title: A Real World, Observational Pediatric Registry of the Acclarent AERA® Eustachian Tube Balloon Dilation System
Brief Title: AERA Pediatrics Registry
Status: Recruiting | Type: Observational
Sponsor: Integra LifeSciences Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: C-AERA-P-001
Record Dates: First submitted 2025-07-08; First posted 2025-07-17 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Dysfunction of Eustachian Tube
Keywords: ETBD

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 27 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Prospective, multi-center, observational, real-world evidence data collection registry to confirm the continued clinical performance of the AERA® device in pediatric patients

ELIGIBILITY:
Inclusion Criteria:

1. Age <18
2. Specific indications for ETBD are documented
3. ETBD with AERA device attempted-

Exclusion Criteria:

1. ETBD with device other than AERA®
2. Previous ETBD procedure-

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects under the age of 18 with ETD who are treated with the AERA® device
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-06-17 (Actual); Primary Completion 2030-10 (Estimated); Study Completion 2031-02 (Estimated)

PRIMARY OUTCOMES:
Failure-free after ETBD with the AERA® device. | 27 months
  Failure is defined as revision ETD surgery (e.g. further ETBD, tympanostomy tube (TT) insertion, or adenoidectomy for ETD).

SECONDARY OUTCOMES:
Tympanogram assessed by ear | 27 months
  Tympanogram
Pure tone audiometry (PTA) assessed by ear | 27 months
  Pure tone audiometry (PTA)
Valsalva maneuver assessed by ear | 27 months
  Valsalva maneuver
Inflammation score assessed by ear | 27 months
  Score 1-4. The higher the score, the worse the outcome.
Eustachian Tube Dysfunction Questionnaire (ETDQ-7) assessed by patient | 27 months
  Total score of 7-49. The higher the score, the worse the outcome.
Otitis Media- 6 Questionnaire (OM-6) assessed by patient | 27 months
  Total score 6-42. The higher the score, the worse the outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Schutt, MD, Study Director — Acclarent, an Integra LifeSciences Company
Locations (6):
- United States (6):
  - Stanford University, Palo Alto, California
  - Michigan Pediatric ENT Associates, West Bloomfield, Michigan
  - Children's Minnesota, Minneapolis, Minnesota
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Ear and Sinus Institute, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: Undecided